CLINICAL TRIAL: NCT01315561
Title: Motion Style Acupuncture Treatment for Low Back Pain With Severe Disability: a Randomised, Controlled, Trial Protocol
Brief Title: Motion Style Acupuncture Treatment for Low Back Pain With Severe Disability
Acronym: MSAT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jaseng Hospital of Korean Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JSR-2011-01
Record Dates: First submitted 2011-03-14; First posted 2011-03-15 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Complete Immobility Due to Severe Physical Disability
Keywords: acute low back pain; motion stlye acupuncture treatment; disability; MSAT
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- acupuncture (Experimental): MSAT is a treatment method in which the patient is exposed to active or passive movement and exercise during acupuncture, as opposed to conventional acupuncture.
  Interventions: Other: acupuncture, injection
- injections of diclofenac (Active Comparator): the control group was treated with intramuscular injections of diclofenac(NSAID). All administrations were limited to 1 session
  Interventions: Other: acupuncture, injection

INTERVENTIONS:
Other: acupuncture, injection — MSAT and intramuscular injections of diclofenac(NSAID)

SUMMARY:
Motion style acupuncture treatment(MSAT) is a treatment method in which the patient is exposed to active or passive movement and exercise during acupuncture, as opposed to conventional acupuncture. The purpose of this study is to investigate the effect of MSAT in the treating pain and severe functional disability in acute LBP patients.

DETAILED DESCRIPTION:
58 patients with acute LBP and severe disability with an Oswestry Disability Index(ODI) of 60% or higher were randomly allocated and divided into 2 groups. The experimental group was treated with MSAT and the control group was treated with intramuscular injections of diclofenac(NSAID). All administrations were limited to 1 session, and comparisons were made of measurements before and after treatment. Primary outcomes were measured by the NRS(numerical rating scale) of back pain in active movement. Secondary outcomes were measured by the NRS of radiating pain, ODI scores, and the patient's global impression of change(PGIC) etc. Post-treatment follow-up will be performed to measure primary and secondary outcomes with the exception of ROM and SLR at 2, 4, and 24 weeks after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Acute LBP(with or without leg pain), with onset within past 4 weeks
* Severe disability as assessed by an Oswestry Disability Index of 60% or higher
* Age between 20 and 60
* Given consent to lumbar MRI
* Voluntary participation with written consent given to study consent form

Exclusion Criteria:

* Diagnosis of serious disease(s) which are possible causes of back pain such as malignancy, vertebral fracture, spinal infection, inflammatory spondylitis, cauda equina compression, etc.
* Prior diagnosis of other chronic disease(s) which could affect effectiveness or interpretation of treatment results such as cardiovascular disease, diabetic neuropathy, fibromyalgia, rheumatoid arthritis, Alzheimer's disease, epilepsy, etc.
* Progressive neurologic deficit(s) or concurrent severe neurological symptoms
* Unsuitable for or at risk of complications from acupuncture treatment such as patients with clotting disorders, severe diabetes with risk of infection, serious cardiovascular disease, or undergoing anticoagulant treatment, etc.
* Under prescription of corticosteroids, immuno-suppressant drugs, psychiatric medicine, or other medication considered unsuitable for subjects by the researcher
* Experience of gastroenteric complications after taking NSAIDs or currently undergoing treatment for digestive disorders
* During pregnancy or suspected pregnancy
* Subjects considered unsuitable for clinical trial by the researcher

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2011-10 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in numerical rating scale of back pain | Before treatment, At 30 minutes, 2, 4, and 24 weeks after treatment.

SECONDARY OUTCOMES:
Change from Baseline in NRS of radiating pain, ODI scores, and the patient's global impression of change(PGIC),range of motion (ROM) of the lumbar spine, and degrees of straight leg raising (SLR) | Before treatment, At 30 minutes, 2, 4, and 24 weeks after treatment.
  Post-treatment follow-up will be performed to measure primary and secondary outcomes with the exception of ROM and SLR at 2, 4, and 24 weeks after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Joonshik Shin, Principal Investigator — JASENG HOSPITAL
Locations (2):
- South Korea (2):
  - Jaseng Oriental Hospital, Seoul, Gangnamgu Sinsadong
  - Jaseng Oriental Hospital, Bucheon-si

REFERENCES:
- [Derived] Shin JS, Ha IH, Lee TG, Choi Y, Park BY, Kim MR, Lee MS. Motion style acupuncture treatment (MSAT) for acute low back pain with severe disability: a multicenter, randomized, controlled trial protocol. BMC Complement Altern Med. 2011 Dec 13;11:127. doi: 10.1186/1472-6882-11-127. PMID 22151475